CLINICAL TRIAL: NCT05079750
Title: A Phase I Study to Determine the Safety and Immunogenicity of a Bivalent ChAdOx1 Vectored Vaccine Against Zaire and Sudan Ebola Virus Species in UK Healthy Adult Volunteers
Brief Title: A Study of a New Vaccine Against Two Types of Ebola
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: EBL07
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2021-10

CONDITIONS: Ebola
Keywords: Ebola Virus Disease; Zaire Ebolavirus; EBOV; Sudan Ebolavirus; SUDV; Vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Low Dose (Experimental): n=6 participants vaccinated with a single dose of ChAdOx1 biEBOV 5x10^9 vp
  Interventions: Biological: ChAdOx1 biEBOV
- Group 2: Mid Dose (Experimental): n=6 participants vaccinated with a single dose of ChAdOx1 biEBOV 2.5x10^10 vp
  Interventions: Biological: ChAdOx1 biEBOV
- Group 3: High Dose (Experimental): n=14 participants vaccinated with either a single dose (n=7) or two doses twelve weeks apart (n=7) of ChAdOx1 biEBOV 5x10^10 vp
  Interventions: Biological: ChAdOx1 biEBOV

INTERVENTIONS:
Biological: ChAdOx1 biEBOV — ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)

SUMMARY:
An open-label, non-randomised, dose escalation, first-in-human, single centre, phase I clinical trial to determine the safety and immunogenicity of a bivalent ChAdOx1 vectored vaccine against Zaire and Sudan Ebola virus species in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, dose escalation, phase I clinical trial to assess the safety and immunogenicity of the candidate ChAdOx1 biEBOV vaccine in healthy UK volunteers aged 18-55. The vaccine will be administered intramuscularly (IM).

Volunteers will be recruited and vaccinated at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford. There will be 3 study groups and it is anticipated that a total of 26 volunteers will be enrolled. Dose escalation and sentinel participant procedures will be implemented. Volunteers will be first recruited into Group 1 and subsequently into Groups 2 and 3 following interim clinical safety reviews. Volunteers will be sequentially allocated to a study group by selecting eligible volunteers for enrolment following screening. Sequential allocation will occur based on the order in which volunteers are enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 55 years.
2. Able and willing (in the Investigator's opinion) to comply with all study requirements.
3. Willing to allow confirmation of their past medical history either through: provision of a GP medical record summary, allowing investigators to obtain a copy of their medical history from their GP practice or by providing an alternative acceptable means of confirming their past medical history.
4. Agreement to refrain from blood donation during the course of the study.
5. Provide written informed consent.
6. For women of childbearing potential only: Willingness to practice continuous effective contraception for the duration of the trial.
7. For women of childbearing potential only: A negative pregnancy test on the day of both screening and vaccination.

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period.
2. Receipt of a recombinant simian adenoviral vaccine prior to enrolment.
3. Planned receipt of another adenoviral vectored vaccine (e.g. Oxford/AstraZeneca or Janssen COVID-19 vaccines) within 90 days after the vaccination with the ChAdOx1 biEBOV.
4. Planned or actual receipt of any vaccines administered within 30 days (before or after) enrolment and/or planned receipt of a vaccine ≤30 days after enrolment EXCEPT for protein, RNA (or other non-adenovirus based) COVID-19 vaccinations which may be given within 14 days of the trial vaccine.
5. Previous receipt of an Ebolavirus vaccine.
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
7. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) systemically active immunosuppressant medication within the past 6 months.
8. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Including hypersensitivity to the active substance or to any of the excipients of the IMP or Vaxzevria (i.e. the Oxford/AstraZeneca COVID-19 vaccine).
9. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
10. History of anaphylaxis in relation to vaccination.
11. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
12. History of serious psychiatric condition likely to affect participation in the study.
13. Ongoing or planned pregnancy or breastfeeding during the trial follow up period.
14. Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
15. History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), history of antiphospholipid syndrome, or history of heparin induced thrombocytopenia.
16. Individuals who have experienced thrombosis with thrombocytopenia syndrome (TTS) following vaccination with Vaxzevria (i.e. the Oxford/AstraZeneca COVID-19 vaccine).
17. Individuals who have previously experienced episodes of capillary leak syndrome.
18. Any other serious chronic illness requiring hospital specialist supervision.
19. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
20. Suspected or known injecting drug abuse in the 5 years preceding enrolment.
21. Detectable circulating hepatitis B surface antigen (HBsAg).
22. Seropositive for hepatitis C virus (antibodies to HCV).
23. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
24. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cicconi, Dr., Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkin D, Makinson R, Sanders H, Sampson A, Platt A, Tran N, Dinesh T, Mabbett R, Lawrie A, Quaddy J, Poulton I, Berrie E, Cicconi P, Lambe T. Safety and immunogenicity of a bivalent Ebola virus and Sudan virus ChAdOx1 vectored vaccine in adults in the UK: an open-label, non-randomised, first-in-human, phase 1 clinical trial. Lancet Microbe. 2025 May;6(5):101022. doi: 10.1016/j.lanmic.2024.101022. Epub 2025 Feb 5. PMID 39922207

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose
Started | 6 | 6 | 14
Completed | 6 | 6 | 13 (Participant who received a single high dose of vaccine was lost to follow-up after attending the D28 visit)
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 3: High Dose - Single Dose: n=7 participants vaccinated with a single dose of ChAdOx1 biEBOV 5x10^10 vp
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
- Group 3: High Dose - Two Doses: n=7 participants vaccinated with two doses twelve weeks apart of ChAdOx1 biEBOV 5x10^10 vp
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
- Total: Total of all reporting groups
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 26
Age, Customized [Median (Inter-Quartile Range); unit: years] | 24 [19 to 31] | 26 [22 to 32] | 20 [19 to 28] | 30 [28 to 33] | 28 [20 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 4 | 16
  Male | 2 | 3 | 2 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 4 | 4 | 7 | 21
  Black Carribean and Mixed White or | 0 | 1 | 0 | 0 | 1
  Asian or Asian British | 0 | 0 | 2 | 0 | 2
  Other Asian Background | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6 | 6 | 7 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of ChAdOx1 biEBOV in Healthy Volunteers: Number of Participants With Occurrence of Solicited Local and Systemic Reactogenicity Signs and Symptoms
Description: Occurrence of solicited local and systemic reactogenicity signs and symptoms. Data shown are number (and percentage) of participants reporting each event. The maximum severity of any local and any systemic solicited symptoms reported by individual participants is also shown.
Time Frame: 7 days following vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: High Dose - Single Dose: n=14 participants vaccinated with dose 1 of ChAdOx1 biEBOV 5x10^10 vp
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
- Group 3: High Dose - Two Doses: n=7 participants vaccinated with dose 2 of ChAdOx1 biEBOV 5x10^10 vp
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
Participants
  Any local symptom: Mild | 3 | 3 | 9 | 4
  Any local symptom: Moderate | 0 | 1 | 1 | 1
  Any local symptom: Severe | 0 | 0 | 0 | 0
  Any local symptom: Did not report this event | 3 | 2 | 4 | 2
  Pain: Mild | 3 | 4 | 9 | 4
  Pain: Moderate | 0 | 0 | 1 | 1
  Pain: Severe | 0 | 0 | 0 | 0
  Pain: Did not report this event | 3 | 2 | 4 | 2
  Redness: Mild | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0
  Redness: Did not report this event | 6 | 6 | 14 | 7
  Itch: Mild | 1 | 1 | 0 | 0
  Itch: Moderate | 0 | 0 | 0 | 0
  Itch: Severe | 0 | 0 | 0 | 0
  Itch: Did not report this event | 5 | 5 | 14 | 7
  Warmth: Mild | 2 | 1 | 2 | 1
  Warmth: Moderate | 0 | 1 | 0 | 0
  Warmth: Severe | 0 | 0 | 0 | 0
  Warmth: Did not report this event | 4 | 4 | 12 | 6
  Any systemic symptom: Mild | 3 | 3 | 2 | 2
  Any systemic symptom: Moderate | 3 | 2 | 10 | 3
  Any systemic symptom: Severe | 0 | 0 | 0 | 0
  Any systemic symptom: Did not report this event | 0 | 1 | 2 | 2
  Fever: Mild | 0 | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0 | 1
  Fever: Severe | 0 | 0 | 0 | 0
  Fever: Did not report this event | 6 | 6 | 14 | 6
  Myalgia: Mild | 0 | 2 | 6 | 2
  Myalgia: Moderate | 0 | 0 | 4 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Did not report this event | 6 | 4 | 4 | 5
  Nausea: Mild | 3 | 1 | 4 | 1
  Nausea: Moderate | 0 | 0 | 1 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Did not report this event | 3 | 5 | 9 | 6
  Malaise: Mild | 1 | 4 | 4 | 3
  Malaise: Moderate | 0 | 0 | 6 | 1
  Malaise: Severe | 0 | 0 | 0 | 0
  Malaise: Did not report this event | 5 | 2 | 4 | 3
  Arthralgia: Mild | 1 | 2 | 1 | 1
  Arthralgia: Moderate | 0 | 0 | 3 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Did not report this event | 5 | 4 | 10 | 6
  Fatigue: Mild | 2 | 3 | 6 | 0
  Fatigue: Moderate | 2 | 1 | 5 | 3
  Fatigue: Severe | 0 | 0 | 0 | 0
  Fatigue: Did not report this event | 2 | 2 | 3 | 4
  Feverishness: Mild | 2 | 0 | 6 | 1
  Feverishness: Moderate | 0 | 1 | 4 | 0
  Feverishness: Severe | 0 | 0 | 0 | 0
  Feverishness: Did not report this event | 4 | 5 | 4 | 6
  Headache: Mild | 3 | 3 | 6 | 3
  Headache: Moderate | 1 | 1 | 4 | 1
  Headache: Severe | 0 | 0 | 0 | 0
  Headache: Did not report this event | 2 | 2 | 4 | 3

2. Primary Outcome: Safety and Tolerability of ChAdOx1 biEBOV in Healthy Volunteers: Number of Participants With Occurrence of Unsolicited Signs and Symptoms
Description: Occurrence of unsolicited adverse events (AEs)
Time Frame: 28 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
Participants
  Cardiac disorders (vaccine-related) | 0 | 2 | 0 | 0
  Gastrointestinal disorders (vaccine-related) | 1 | 1 | 1 | 0
  General disorders and administration site reactions (vaccine-related) | 0 | 2 | 2 | 1
  Musculoskeletal and connective tissue disorders (vaccine-related) | 0 | 0 | 3 | 0
  Infections and infestations (vaccine-related) | 0 | 0 | 0 | 1
  Nervous system disorders (vaccine-related) | 0 | 1 | 3 | 0
  Reproductive system and breast disorders (vaccine-related) | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders (vaccine-related) | 2 | 2 | 1 | 2
  Cardiac disorders (vaccine-unrelated) | 0 | 0 | 0 | 0
  Gastrointestinal disorders (vaccine-unrelated) | 3 | 0 | 1 | 3
  General disorders and administration site reactions (vaccine-unrelated) | 3 | 0 | 3 | 2
  Musculoskeletal and connective tissue disorders (vaccine-unrelated) | 1 | 0 | 1 | 0
  Infections and infestations (vaccine-unrelated) | 0 | 1 | 0 | 3
  Nervous system disorders (vaccine-unrelated) | 1 | 2 | 3 | 3
  Reproductive system and breast disorders (vaccine-unrelated) | 1 | 1 | 0 | 0
  Respiratory, thoracic and mediastinal disorders (vaccine-unrelated) | 1 | 2 | 5 | 4

3. Primary Outcome: Safety and Tolerability of ChAdOx1 biEBOV in Healthy Volunteers: Number of Participants With Occurrence of Serious Adverse Events
Description: Occurrence of serious adverse events (SAEs) and adverse interests of special interest (AESIs)
Time Frame: Duration of the study (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
Participants | 1 | 0 | 0 | 0

4. Primary Outcome: Safety and Tolerability of ChAdOx1 biEBOV in Healthy Volunteers: Number of Participants With Occurrence of Clinical Laboratory Abnormalities
Description: Abnormal results were graded according to a pre-specified laboratory adverse events severity grading scale - a full breakdown of the levels of severity of the reported events per study timepoint is available in the publication.
Time Frame: 28 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
Participants
  Alanine transaminase: Normal | 6 | 5 | 14 | 7
  Alanine transaminase: Abnormal | 0 | 1 | 0 | 0
  Albumin: Normal | 5 | 6 | 14 | 7
  Albumin: Abnormal | 1 | 0 | 0 | 0
  Alkaline phosphatase: Normal | 6 | 6 | 14 | 7
  Alkaline phosphatase: Abnormal | 0 | 0 | 0 | 0
  Bilirubin: Normal | 5 | 5 | 10 | 5
  Bilirubin: Abnormal | 1 | 1 | 4 | 2
  Creatinine: Normal | 6 | 6 | 14 | 7
  Creatinine: Abnormal | 0 | 0 | 0 | 0
  Potassium: Normal | 6 | 6 | 10 | 5
  Potassium: Abnormal | 0 | 0 | 4 | 2
  Sodium: Normal | 6 | 6 | 14 | 7
  Sodium: Abnormal | 0 | 0 | 0 | 0
  Urea: Normal | 6 | 6 | 14 | 7
  Urea: Abnormal | 0 | 0 | 0 | 0
  Eosinophil count: Normal | 6 | 6 | 14 | 7
  Eosinophil count: Abnormal | 0 | 0 | 0 | 0
  Hemoglobin: Normal | 5 | 6 | 12 | 7
  Hemoglobin: Abnormal | 1 | 0 | 2 | 0
  Lymphocyte count: Normal | 5 | 4 | 6 | 7
  Lymphocyte count: Abnormal | 1 | 2 | 8 | 0
  Neutrophil count: Normal | 6 | 4 | 9 | 5
  Neutrophil count: Abnormal | 0 | 2 | 5 | 2
  Platelet count: Normal | 6 | 6 | 13 | 6
  Platelet count: Abnormal | 0 | 0 | 1 | 1
  White blood cell count: Normal | 6 | 5 | 14 | 7
  White blood cell count: Abnormal | 0 | 1 | 0 | 0

5. Secondary Outcome: Immunogenicity of ChAdOx1 biEBOV in Healthy Adult Volunteers: Measure of Humoral Immunogenicity
Description: ELISA to quantify antibodies to filovirus glycoprotein (specific serological response). Peak antibody responses to both Ebola and Sudan viruses occurred 28 days post vaccination (or post-boost, in the participants who received a booster) across all groups.
Time Frame: At day 28
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
ELISA units
  Peak anti-EBOV antibody titers (occurred at D28) | 63.3 [7.2 to 555.0] | 164.2 [88.9 to 303.1] | 260.1 [132.9 to 509.1] | 1169.7 [719.8 to 1902.5]
  Peak anti-SUDV antibody titers (occurred at D28) | 27.0 [4.9 to 148.5] | 101.7 [48.4 to 213.8] | 111.5 [48.2 to 256.6] | 568.0 [296.4 to 1088]

6. Secondary Outcome: Immunogenicity of ChAdOx1 biEBOV in Healthy Adult Volunteers: Measure of Cellular Immunogenicity
Description: Intracellular cytokine staining (ICS) by flow cytometry was carried out at baseline as well as at 14 days after vaccination/boost to assess T-cell responses to Ebola virus glycoprotein and Sudan virus glycoprotein.
Time Frame: 14 days post final vaccine for each group
Measure: Median (Inter-Quartile Range); unit: frequency (proportion of parent cells)
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose - Single Dose | Group 3: High Dose - Two Doses
Number analyzed (Participants) | 6 | 6 | 14 | 7
frequency (proportion of parent cells)
  Antigen-specific CD8+ T cells to EBOV | 0.0300 [0.0090 to 0.0395] | 0.0000 [0.0000 to 0.6945] | 0.0850 [0.0010 to 0.2075] | 0.1190 [0.0000 to 0.3553]
  Antigen-specific CD8+ T cells to SUDV | 0.0320 [0.0150 to 0.0665] | 0.0340 [0.0000 to 0.5415] | 0.1120 [0.0425 to 0.3495] | 0.0485 [0.0188 to 0.4538]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs were collected 7 days post each vaccination. Unsolicited adverse events were collected 28 days post each vaccination. Serious adverse events and adverse events of special interest were collected for each volunteer from their enrolment to their final visit.
Groups:
- Group 3: High Dose 1: n=14 participants vaccinated with a single dose of ChAdOx1 biEBOV 5x10^10 vp
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
- Group 4: High Dose 2: n=7 participants vaccinated with a second dose of ChAdOx1 biEBOV 5x10^10 vp twelve weeks after the first
  ChAdOx1 biEBOV: ChAdOx1 biEBOV provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: High Dose 1 | Group 4: High Dose 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 12/14 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Low Dose (N=6) | Group 2: Mid Dose (N=6) | Group 3: High Dose 1 (N=14) | Group 4: High Dose 2 (N=7)
Endometriotic cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to the vaccine. Classified as an SAE since it led to hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Low Dose (N=6) | Group 2: Mid Dose (N=6) | Group 3: High Dose 1 (N=14) | Group 4: High Dose 2 (N=7)
Solicited local AEs (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 10 (10) | 5 (5) — Listed in detail in Outcome Measure 1
Solicited systemic AEs (Immune system disorders) | 6 (6) | 5 (5) | 12 (12) | 5 (5) — Listed in detail in Outcome Measure 1
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ucler (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (2) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hordoleum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site dryness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased viscosity of upper respiratory tract (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT05079750/Prot_SAP_000.pdf